CLINICAL TRIAL: NCT04420975
Title: A Phase I Study of Nivolumab and Intratumoral BO 112 for Resectable Soft Tissue Sarcoma
Brief Title: Nivolumab and BO-112 Before Surgery for the Treatment of Resectable Soft Tissue Sarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Highlight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-000419; NCI-2019-08556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1K08CA245181-01 (NIH)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Leiomyosarcoma; Malignant Peripheral Nerve Sheath Tumor; Myxofibrosarcoma; Pleomorphic Rhabdomyosarcoma; Resectable Dedifferentiated Liposarcoma; Resectable Soft Tissue Sarcoma; Resectable Undifferentiated Pleomorphic Sarcoma; Soft Tissue Fibrosarcoma; Spindle Cell Sarcoma; Stage I Retroperitoneal Sarcoma AJCC (American Joint Committee on Cancer) v8; Stage I Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IA Retroperitoneal Sarcoma AJCC v8; Stage IA Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IB Retroperitoneal Sarcoma AJCC v8; Stage IB Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage II Retroperitoneal Sarcoma AJCC v8; Stage II Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage III Retroperitoneal Sarcoma AJCC v8; Stage III Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIA Retroperitoneal Sarcoma AJCC v8; Stage IIIA Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIB Retroperitoneal Sarcoma AJCC v8; Stage IIIB Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Storiform-Pleomorphic Malignant Fibrous Histiocytoma; Synovial Sarcoma; Undifferentiated High Grade Pleomorphic Sarcoma of Bone; Undifferentiated Pleomorphic Sarcoma; Undifferentiated Pleomorphic Sarcoma With Osteoclast-Like Giant Cells; Undifferentiated Pleomorphic Sarcoma, Inflammatory Variant; Undifferentiated Spindle Cell Sarcoma
MeSH Terms: conditions — Leiomyosarcoma; Neurofibrosarcoma; Dermatofibrosarcoma; Sarcoma; Histiocytoma, Malignant Fibrous; Sarcoma, Synovial | interventions — BO-112; Nivolumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (BO-112, nivolumab) (Experimental): Patients receive BO-112 intratumorally on days 8 and 15 or 1, 8, and 15 and nivolumab IV over 30-60 minutes on day 8 in the absence of disease progression or unacceptable toxicity. Patients also undergo standard of care radiation therapy on days 8-12 for a total of 5 fractions. Patients then undergo standard of care definitive surgical resection on day 26 to 50.
  Interventions: Procedure: Definitive Surgical Resection; Biological: Nanoplexed Poly I:C BO-112; Biological: Nivolumab; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Definitive Surgical Resection — Undergo definitive surgical resection
Biological: Nanoplexed Poly I:C BO-112 — Given intratumorally
  Other Names: BO 112; BO-112; BO112; Nanoplexed Poly IC BO-112; Nanoplexed Polyinosinic:Polycytidylic Acid BO-112
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects of BO-112 when given together with nivolumab before surgery in treating patients with soft tissue sarcoma that can be removed by surgery (resectable). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Immunotherapy with BO-112, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving nivolumab and BO-112 before surgery may work better in treating patients with soft tissue sarcoma compared to nivolumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of integrating BO-112, and BO-112 with nivolumab in soft tissue sarcoma patients undergoing preoperative radiotherapy.

SECONDARY OBJECTIVES:

I. Determine the change in T cell infiltration at surgical resection from baseline as measured by immunohistochemistry.

II. Assess treatment effect (necrosis score) of BO-112 and BO-112 in combination with nivolumab in soft tissue sarcoma patients receiving preoperative hypofractionated radiotherapy, compared to patients treated on a recently completed phase 2 study of preoperative hypofractionated radiotherapy alone.

III. Evaluate the 2-year rate of local and distant metastasis of BO-112 and BO-112 in combination with nivolumab in patients with localized resectable soft tissue sarcoma receiving preoperative hypofractionated radiotherapy, as compared to historical patients receiving preoperative radiotherapy alone.

EXPLORATORY OBJECTIVES:

I. Evaluate the dynamics of the intratumoral T cell phenotype. II. Assess the capacity to grow ex vivo tumor infiltrating lymphocytes from patients treated with BO-112 and BO-112 in combination with nivolumab.

III. Analyze changes in T-cell receptor (TCR) repertoire in tumor infiltrating lymphocytes and peripheral blood mononuclear cells (PBMCs) between baseline, post-treatment, and ex vivo cultured tumor infiltrating lymphocyte (TIL) samples.

IV. For patients with disease burden outside of the resected lesion, assess imaging response to treatment using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

OUTLINE:

Patients receive BO-112 intratumorally on days 8 and 15 or 1, 8, and 15 and nivolumab intravenously (IV) over 30-60 minutes on day 8 in the absence of disease progression or unacceptable toxicity. Patients also undergo standard of care radiation therapy on days 8-12 for a total of 5 fractions. Patients then undergo standard of care definitive surgical resection on day 26 to 50.

After completion of study treatment, patients are followed up at 2 weeks, 3 months, and between 6-12, 12-18, and 18-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, and assent where appropriate, must be obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Biopsy proven soft tissue sarcoma of the extremity, trunk or retroperitoneum including undifferentiated pleomorphic sarcoma, myxofibrosarcoma, leiomyosarcoma, dedifferentiated liposarcoma, synovial sarcoma, malignant peripheral nerve sheath tumor, or pleomorphic rhabdomyosarcoma. Undifferentiated pleomorphic sarcoma encompasses any of the following histologies:

  * Pleomorphic undifferentiated sarcoma
  * Unclassified spindle cell sarcoma
  * Spindle cell sarcoma not otherwise specified
  * Pleomorphic spindle cell sarcoma
  * Pleomorphic fibroblastic sarcoma
  * Undifferentiated high-grade pleomorphic sarcoma
  * Pleomorphic sarcoma with prominent inflammation
  * Pleomorphic sarcoma with giant cells
  * Malignant fibrous histiocytoma (including storiform-pleomorphic and inflammatory subtypes)
  * Fibrosarcoma
* Tumor that is injectable
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 100,000/mm^3 and transfusion independent
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (ULN)
* Serum creatinine < 1.5 x ULN or creatinine clearance > 60 mL/min for patients with creatinine levels above ULN (as determined by Cockcroft-Gault equation)
* Bilirubin =< 1.5 x ULN; for subjects with documented/suspected Gilbert's disease, bilirubin =< 3 x ULN
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal unless the patient is on anticoagulant therapy within 28 days prior to enrollment (if the patient is receiving anticoagulant therapy, PT, and a PTT must be within therapeutic range of intended use of anticoagulants)
* Patients must be willing to submit blood and tissue specimens for translational medicine studies
* Patients must be offered the opportunity to participate in specimen banking for future research
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug
* Women must not be breastfeeding
* Women of childbearing potential (WOCBP) must be willing to use either two adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy, or to abstain from heterosexual activity (complete abstinence) throughout the study, starting with visit 1 through 5 months after the last dose of study therapy. Approved contraceptive methods include intrauterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, female condoms with spermicide, or oral contraceptives. Spermicides alone are not an acceptable method of contraception. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to highly effective contraception during active participation in study treatment and for a period of 7 months after the last dose of nivolumab
* HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly. WOCBP and female partners of male subjects, who are WOCBP, are expected to use one of the highly effective methods of contraception listed below. Male subjects must inform their female partners who are WOCBP of the contraceptive requirements of the protocol and are expected to adhere to using contraception with their partner. Contraception methods are as follows:

* Progestogen only hormonal contraception associated with inhibition of ovulation
* Hormonal methods of contraception including oral contraceptive pills containing combined estrogen + progesterone, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena
* Nonhormonal IUDs, such as ParaGard
* Bilateral tubal occlusion
* Vasectomized partner with documented azoospermia 90 days after procedure

  * Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success
* Intrauterine hormone-releasing system (IUS)
* Complete abstinence

  * Complete abstinence is defined as the complete avoidance of heterosexual intercourse
  * Complete abstinence is an acceptable form of contraception for all study drugs and must be used throughout the duration of the study treatment (plus 5 half-lives of the investigational drug plus 30 days)
  * It is not necessary to use any other method of contraception when complete abstinence is elected
  * Subjects who choose complete abstinence must continue to have pregnancy tests, as specified
  * Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence
  * The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject

    * LESS EFFECTIVE METHODS OF CONTRACEPTION
* Diaphragm with spermicide
* Cervical cap with spermicide
* Vaginal sponge with spermicide
* Male or female condom with or without spermicide

  * A male and a female condom must not be used together
* Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action

  * UNACCEPTABLE METHODS OF CONTRACEPTION
* Periodic abstinence (calendar, symptothermal, post-ovulation methods)
* Withdrawal (coitus interruptus)
* Spermicide only
* Lactation amenorrhea method (LAM)

Exclusion Criteria:

* Contraindications to tumor biopsy and injections (coagulopathy, known history of keloid formation, etc.)
* Women who are pregnant or breastfeeding
* Inability to give informed consent
* History of other malignancy that can interfere with interpretation of the results
* Prior irradiation in the area to be treated with preoperative radiation such that the risk of re-irradiation outweighs its benefit, according to the treating radiation oncologist
* Any condition that might interfere with the subject's participation in the study, safety, or in the evaluation of the study results
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
* Patients must not have received any live vaccine within 30 days prior to registration. Seasonal flu vaccines and other vaccines that do not contain live virus are permitted
* Any concurrent chemotherapy, immunotherapy, or biologic therapy for cancer treatment. Concurrent use of hormones is acceptable
* Patient must not have evidence of any clinically significant immunosuppression such as the following: primary immunodeficiency state such as severe combined immunodeficiency disease; concurrent opportunistic infection; receiving systemic immunosuppressive therapy within 28 days before enrollment with the exceptions of intranasal, topical, and inhaled corticosteroids or oral corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
* Active or prior documented autoimmune disease within the past 3 years

  * NOTE: Subjects with active, known or suspected autoimmune disease such as vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Active or prior documented inflammatory bowel disease
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids or has current ILD/pneumonitis or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Current or history of fibromyalgia, myositis, myocarditis or myasthenia gravis
* Exposure to any investigational drug within 7 days prior to screening visit or for which 5 half-lives have not elapsed
* Prisoners or subjects who are involuntarily incarcerated

  * Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a subject
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | study enrollment through 100 days after the last dose of study drug
  AEs will be tabulated by type, severity, and the proportion of subject experiencing the event.

SECONDARY OUTCOMES:
Immune-oncologic impact of the BO-112 or the combined regimen of nivolumab and BO-112 | from the date of study drug initiation until 50 days after study drug initiation (or the date of surgery, whichever comes first)
  Statistical analysis of immune-oncologic changes will be performed by comparing results from surgical specimens with baseline biopsy specimens. For immunohistochemical parameters, the percentage of CD4+ (cluster of differentiation 4) or CD8+((cluster of differentiation 8) cells will be compared between biopsy and surgical specimens using a paired two-tailed ratio T-test comparing means.
Pathologic treatment effect | At time of surgery
  Will be compared to historical samples receiving preoperative radiotherapy alone. Will use a two-sample paired T-test comparing means.

CONTACTS AND LOCATIONS:
Overall Officials: Vishruth Reddy, MD, PhD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States